CLINICAL TRIAL: NCT05243342
Title: A Phase Ib, Open-Label, Multicenter, Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of XMAB24306 in Combination With Daratumumab in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of XMAB24306 in Combination With Daratumumab in Participants With Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO43073
Record Dates: First submitted 2022-02-01; First posted 2022-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation (Experimental): Participants will receive escalating doses of XmAb24306 with daratumumab up to the maximum tolerated dose (MTD)
  Interventions: Drug: XmAb24306; Drug: Daratumumab
- Dose expansion (Experimental): Participants will receive XmAb24306 with daratumumab at the recommended phase 2 dose (RP2D)
  Interventions: Drug: XmAb24306; Drug: Daratumumab

INTERVENTIONS:
Drug: XmAb24306 — XmAb24306 will be given via intravenous (IV) infusion
  Other Names: RO7310729
Drug: Daratumumab — Participants will receive daratumumab via subcutaneous (SC) injection every week for Cycles 1-4, every 2 weeks for Cycles 5-12, and every 4 weeks thereafter (cycle length = 2 weeks for Cycles 1-12 and 4 weeks thereafter)

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics, and activity of XmAb24306 in combination with a multiple myeloma (MM)-targeting monoclonal antibody capable of inducing antibody-dependent cellular toxicity (ADCC) in participants with relapsed or refractory (R/R) MM who have received a minimum of three prior treatments, including at least one immunomodulatory drug (IMiD), one proteasome inhibitor (PI), and one anti-CD38 monoclonal antibody.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* Measurable disease, as defined by the protocol
* Participants must have received a minimum of 3 prior lines of therapy, including at least one PI, one IMiD, and an anti-CD38 monoclonal antibody
* Best response of stable disease or better with at least one prior anti-CD38 monoclonal antibody containing line of treatment

Exclusion Criteria:

* Any anti-cancer therapy within 3 weeks prior to initiation of study treatment, with exceptions defined by the protocol
* Prior allogeneic stem cell or solid organ transplantation
* Autologous stem cell transplantation within 100 days prior to initiation of study treatment
* Significant cardiovascular disease
* Known clinically significant liver disease
* Active or history of autoimmune disease or immune deficiency
* Known active infection requiring IV anti-microbial therapy within 14 days prior to first study drug administration
* Primary or secondary plasma cell leukemia
* Current CNS involvement by MM
* Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with adverse events (AEs) | Up to approximately 3 years

SECONDARY OUTCOMES:
Serum concentration of XmAb24306 | Baseline to approximately 3 years
Objective response rate (ORR) | Baseline to approximately 3 years
Prevalence of XmAb24306 anti-drug antibodies (ADAs) | Baseline to approximately 3 years
Incidence of XmAb24306 ADAs | Baseline to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Alfred Hospital, Melbourne, Victoria
- Denmark (2):
  - Odense Universitetshospital, Odense C, Region Syddanmark
  - Sygehus Lillebælt, Vejle, Vejle, Region Syddanmark
- Oslo Universitetssykehus HF, Oslo, Norway
- Spain (2):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).